CLINICAL TRIAL: NCT05220631
Title: A Technological Intervention to Improve Nutrition Among Older Adult Congregate Meal Participants During COVID-19
Brief Title: Digital Nutrition Intervention for Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at San Antonio (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Older Adult Technology Services (Unknown); City of San Antonio Department of Human Services (Unknown); Agile Analytics, LLC (Unknown)
Responsible Party: Principal Investigator, Sarah Ullevig, Associate Professor, The University of Texas at San Antonio
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-21-241; 1R01NR020303-01 (NIH)
Record Dates: First submitted 2022-01-19; First posted 2022-02-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Nutrition Poor; Physical Inactivity; Social Isolation
Keywords: Technology; Older adult; Nutrition; Food security; Physical activity; Social isolation
MeSH Terms: conditions — Malnutrition; Sedentary Behavior; Social Isolation; Motor Activity

STUDY DESIGN:
Intervention Model Description: This intervention will use a closed-cohort stepped wedge design. In a stepped wedge design, the timing of the intervention is randomized by cluster, with sequential crossover of clusters from control to intervention until all clusters have received the intervention. With this design, each cluster contributes data when they are participating in the intervention and when they are not. This study will be a two-step stepped wedge design; each of the seven targeted centers will then be randomly assigned to one of two cohorts. Participants in Cohort 1 will receive the intervention first. Six months after baseline data have been collected, Cohort 1 participants will finish the intervention and crossover will occur as Cohort 2 participants begin the intervention. At the 12-month time point, the second cohort will complete the intervention. Data will be collected for both groups in each time period T0-T3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will start the intervention directly after randomization.
  Interventions: Behavioral: Technology intervention; Behavioral: Digital Nutrition Intervention
- Cohort 2 (Active Comparator): Cohort 2 will serve as the control while cohort 1 is in the intervention stage. Cohort 2 will start the intervention after cohort 1 concludes the intervention.
  Interventions: Behavioral: Technology intervention; Behavioral: Digital Nutrition Intervention

INTERVENTIONS:
Behavioral: Technology intervention — Older Adult Technology Services (OATS) 5-week technology intervention
Behavioral: Digital Nutrition Intervention — 15-week nutrition intervention delivered completely online

SUMMARY:
The "digital divide" or gap in technological access and knowledge, for older adults has worsened during the COVID-19 pandemic, leading to disruptions in services like congregate meal programs funded by the Older Americans Act. Seven San Antonio congregate meal sites remained partially open biweekly to distribute meals but no longer offer in-person nutrition education, physical activity classes, and social activities. The proposed project will test the efficacy of digital nutrition intervention with at-risk older adults who attend congregate meal center in areas of high poverty and digital exclusion.

The study is uses a stepped-wedge cluster clinical trial. Key community partners with the Department of Health Services Senior Services Division and Older Adult Technology Services (OATS) will participate in the planning phase, research design, and implementation of the study.

The study aims are:

1. To test the impact of a technology-based intervention on the primary outcomes of food security and diet quality;
2. To determine the effect of the intervention on secondary outcomes of technology knowledge and usage, physical activity, and social isolation and loneliness;
3. To examine the long-term impact and sustainability of technology use on food security, diet quality, physical activity, and social isolation.

If successful, the impact of this program could be applied throughout the national OATS network and to similar CMPs to bridge the digital divide beyond the COVID-19 pandemic

DETAILED DESCRIPTION:
This project will target community-dwelling older adults who are "congregate meal" program (CMP) participants living in areas at-risk of the digital divide. The CMP is funded by the Older Americans Act and serves over 2000 San Antonio older adults who live 33% below the poverty level and 18% considered at high nutritional risk. During the pandemic, seven San Antonio sites in areas with high poverty and digital exclusion remain partially open biweekly to distribute meals but did not hold in-person nutrition education, physical activity classes, and social activities. The proposed project extends existing congregate meal programming infrastructure and partnerships with Older Adults Technology Services (OATS), a national leader in creating health service programs focusing on older adults. The goal of the proposed study is to remove the digital barrier to receiving essential, evidence-based nutrition programming online, utilizing OATS' five-week technology "Essential Series," which has successfully educated thousands of older adults nationwide by providing support for technology and internet connectivity.

This proposed nutrition intervention will enrolled congregate meal participants using a stepped-wedge cluster design with two cohorts to allow for sequential intervention enrollment with simultaneous control and intervention data collection timepoints. Key community partners within Department of Health Services Senior Services Division and OATS will participate in the planning phase, research design, and implementation of the study. Feedback from congregate meal participants in focus groups will guide the development of the intervention.

The 20-week intervention will include 5 weeks technology training, including internet access and devices, followed by 15 weeks of a culturally tailored nutrition intervention via online sessions. The study will recruit 440 older adult from seven at-risk congregate meal sites. Data will be collected at baseline (T0), during the online intervention (T1), after the online intervention (T2) and 6 months post-intervention (T3).

The successful outcome of our study will be impactful because of the potential broader application of this program throughout the national OATS network and to similar CMPs to bridge the digital divide through and beyond the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age
* Inadequate or no working technology device (computer, smart-phone, tablet), no or poor internet connectivity at home, or lack of knowledge and usage of technology
* Food insecurity or low diet quality

Exclusion Criteria:

* Blind
* Terminal disease or illness
* Diagnosis of dementia or Alzheimer's disease
* Unable to read or write in English or Spanish

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Diet Quality as measured by the Healthy Eating Index | Change in diet quality from baseline to 3 and 6 months
  Two non-consecutive 24-hour dietary recalls will be collected and the Healthy Index will be calculated to determine diet quality.

SECONDARY OUTCOMES:
Food Security | Change in food security from baseline to 3 and 6 months
  Food security measured by the USDA's US Adult Food Security Survey Module
Physical Activity | Change in physical activity from baseline to 3 and 6 months
  Physical activity measured by the Physical Activity Scale for the Elderly (PASE)
Technology Use and Access | Change in technology use and access from baseline to 3 and 6 months
  Technology use questionnaire from the National Health & Aging Trends Study
Attitudes Towards Technology | Change in attitudes towards technology from baseline to 3 and 6 months
  Adapted from Attitudes Towards Computers Questionnaire (ATCQ)
Social Isolation | Change in social isolation from baseline to 3 and 6 months
  Social isolation measured by The Social Disconnectedness Scale and the Perceived Isolation Scale
Loneliness | Change in loneliness from baseline to 3 and 6 months
  Loneliness assessed by the 3-item UCAL Loneliness Scale
Malnutrition | Change in malnutrition from baseline to 3 and 6 months
  Malnutrition measured by the Mini Nutrition Assessment Short-Form

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Ullevig, PhD, Principal Investigator — University of Texas at San Antonio
Locations (1):
- University of Texas at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after primary and secondary outcome measures has been analyzed and published.
Access Criteria: Data will be made available for research educational purposes.

REFERENCES:
- [Background] Butler MJ, Barrientos RM. The impact of nutrition on COVID-19 susceptibility and long-term consequences. Brain Behav Immun. 2020 Jul;87:53-54. doi: 10.1016/j.bbi.2020.04.040. Epub 2020 Apr 18. PMID 32311498
- [Background] Morley JE, Vellas B. Editorial: COVID-19 and Older Adults. J Nutr Health Aging. 2020;24(4):364-365. doi: 10.1007/s12603-020-1349-9. No abstract available. PMID 32242202
- [Background] Brooke J, Jackson D. Older people and COVID-19: Isolation, risk and ageism. J Clin Nurs. 2020 Jul;29(13-14):2044-2046. doi: 10.1111/jocn.15274. Epub 2020 May 5. No abstract available. PMID 32239784
- [Background] Krendl AC, Perry BL. The Impact of Sheltering in Place During the COVID-19 Pandemic on Older Adults' Social and Mental Well-Being. J Gerontol B Psychol Sci Soc Sci. 2021 Jan 18;76(2):e53-e58. doi: 10.1093/geronb/gbaa110. PMID 32778899
- [Background] Morrow-Howell N, Galucia N, Swinford E. Recovering from the COVID-19 Pandemic: A Focus on Older Adults. J Aging Soc Policy. 2020 Jul-Oct;32(4-5):526-535. doi: 10.1080/08959420.2020.1759758. Epub 2020 Apr 26. PMID 32336225
- [Background] Amarantos E, Martinez A, Dwyer J. Nutrition and quality of life in older adults. J Gerontol A Biol Sci Med Sci. 2001 Oct;56 Spec No 2:54-64. doi: 10.1093/gerona/56.suppl_2.54. PMID 11730238
- [Background] Ettman CK, Abdalla SM, Cohen GH, Sampson L, Vivier PM, Galea S. Prevalence of Depression Symptoms in US Adults Before and During the COVID-19 Pandemic. JAMA Netw Open. 2020 Sep 1;3(9):e2019686. doi: 10.1001/jamanetworkopen.2020.19686. PMID 32876685
- [Background] Parlapani E, Holeva V, Nikopoulou VA, Sereslis K, Athanasiadou M, Godosidis A, Stephanou T, Diakogiannis I. Intolerance of Uncertainty and Loneliness in Older Adults During the COVID-19 Pandemic. Front Psychiatry. 2020 Aug 19;11:842. doi: 10.3389/fpsyt.2020.00842. eCollection 2020. PMID 32973584
- [Background] Naja F, Hamadeh R. Nutrition amid the COVID-19 pandemic: a multi-level framework for action. Eur J Clin Nutr. 2020 Aug;74(8):1117-1121. doi: 10.1038/s41430-020-0634-3. Epub 2020 Apr 20. No abstract available. PMID 32313188
- [Background] Topinkova E. Aging, disability and frailty. Ann Nutr Metab. 2008;52 Suppl 1:6-11. doi: 10.1159/000115340. Epub 2008 Mar 7. PMID 18382070
- [Background] Bollwein J, Volkert D, Diekmann R, Kaiser MJ, Uter W, Vidal K, Sieber CC, Bauer JM. Nutritional status according to the mini nutritional assessment (MNA(R)) and frailty in community dwelling older persons: a close relationship. J Nutr Health Aging. 2013 Apr;17(4):351-6. doi: 10.1007/s12603-013-0034-7. PMID 23538658
- [Background] Trevisan C, Crippa A, Ek S, Welmer AK, Sergi G, Maggi S, Manzato E, Bea JW, Cauley JA, Decullier E, Hirani V, LaMonte MJ, Lewis CE, Schott AM, Orsini N, Rizzuto D. Nutritional Status, Body Mass Index, and the Risk of Falls in Community-Dwelling Older Adults: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2019 May;20(5):569-582.e7. doi: 10.1016/j.jamda.2018.10.027. Epub 2018 Dec 13. PMID 30554987
- [Background] Wei K, Nyunt MSZ, Gao Q, Wee SL, Ng TP. Long-term changes in nutritional status are associated with functional and mortality outcomes among community-living older adults. Nutrition. 2019 Oct;66:180-186. doi: 10.1016/j.nut.2019.05.006. Epub 2019 May 29. PMID 31310959
- [Background] Verlaan S, Ligthart-Melis GC, Wijers SLJ, Cederholm T, Maier AB, de van der Schueren MAE. High Prevalence of Physical Frailty Among Community-Dwelling Malnourished Older Adults-A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2017 May 1;18(5):374-382. doi: 10.1016/j.jamda.2016.12.074. Epub 2017 Feb 24. PMID 28238676
- [Background] Boreskie KF, Hay JL, Duhamel TA. Preventing Frailty Progression during the COVID-19 Pandemic. J Frailty Aging. 2020;9(3):130-131. doi: 10.14283/jfa.2020.29. No abstract available. PMID 32588024
- [Background] de Faria Coelho-Ravagnani C, Corgosinho FC, Sanches FFZ, Prado CMM, Laviano A, Mota JF. Dietary recommendations during the COVID-19 pandemic. Nutr Rev. 2021 Mar 9;79(4):382-393. doi: 10.1093/nutrit/nuaa067. PMID 32653930
- [Background] Saffel-Shrier S, Johnson MA, Francis SL. Position of the Academy of Nutrition and Dietetics and the Society for Nutrition Education and Behavior: Food and Nutrition Programs for Community-Residing Older Adults. J Nutr Educ Behav. 2019 Jul-Aug;51(7):781-797. doi: 10.1016/j.jneb.2019.03.007. Epub 2019 May 16. PMID 31103435
- [Background] Huffman FG, Vaccaro JA, Vieira ER, Zarini GG. Health-Related Characteristics of Older Adults Who Attend Congregate Meal Sites in the United States. Geriatrics (Basel). 2017 Jul 14;2(3):22. doi: 10.3390/geriatrics2030022. PMID 31011032
- [Background] Sahyoun NR, Pratt CA, Anderson A. Evaluation of nutrition education interventions for older adults: a proposed framework. J Am Diet Assoc. 2004 Jan;104(1):58-69. doi: 10.1016/j.jada.2003.10.013. PMID 14702585
- [Background] Bandayrel K, Wong S. Systematic literature review of randomized control trials assessing the effectiveness of nutrition interventions in community-dwelling older adults. J Nutr Educ Behav. 2011 Jul-Aug;43(4):251-62. doi: 10.1016/j.jneb.2010.01.004. Epub 2011 Mar 2. PMID 21371944
- [Background] Neves FJ, Tomita LY, Liu ASLW, Andreoni S, Ramos LR. Educational interventions on nutrition among older adults: A systematic review and meta-analysis of randomized clinical trials. Maturitas. 2020 Jun;136:13-21. doi: 10.1016/j.maturitas.2020.03.003. Epub 2020 Mar 19. PMID 32386661
- [Background] Brewer D, Dickens E, Humphrey A, Stephenson T. Increased Fruit and Vegetable Intake among Older Adults Participating in Kentucky's Congregate Meal Site Program. Educ Gerontol. 2016;42(11):771-784. doi: 10.1080/03601277.2016.1231511. Epub 2016 Sep 3. PMID 28642630
- [Background] Hersey JC, Cates SC, Blitstein JL, Kosa KM, Santiago Rivera OJ, Contreras DA, Long VA, Singh A, Berman DA. Eat Smart, Live Strong intervention increases fruit and vegetable consumption among low-income older adults. J Nutr Gerontol Geriatr. 2015;34(1):66-80. doi: 10.1080/21551197.2015.1007199. PMID 25803605
- [Background] Wunderlich S, Bai Y, Piemonte J. Nutrition risk factors among home delivered and congregate meal participants: need for enhancement of nutrition education and counseling among home delivered meal participants. J Nutr Health Aging. 2011 Nov;15(9):768-73. doi: 10.1007/s12603-011-0090-9. PMID 22089226
- [Background] van Doorn-van Atten MN, de Groot LC, Romea AC, Schwartz S, de Vries JH, Haveman-Nies A. Implementation of a multicomponent telemonitoring intervention to improve nutritional status of community-dwelling older adults: a process evaluation. Public Health Nutr. 2019 Feb;22(2):363-374. doi: 10.1017/S1368980018002185. Epub 2018 Sep 3. PMID 30175698
- [Background] Mitchell RE, Ash SL, McClelland JW. Nutrition education among low-income older adults: a randomized intervention trial in Congregate Nutrition sites. Health Educ Behav. 2006 Jun;33(3):374-92. doi: 10.1177/1090198105276212. PMID 16699126
- [Background] van Doorn-van Atten MN, Haveman-Nies A, van Bakel MM, Ferry M, Franco M, de Groot LCPGM, de Vries JHM. Effects of a multi-component nutritional telemonitoring intervention on nutritional status, diet quality, physical functioning and quality of life of community-dwelling older adults. Br J Nutr. 2018 May;119(10):1185-1194. doi: 10.1017/S0007114518000843. PMID 29759110
- [Background] Marx W, Kelly JT, Crichton M, Craven D, Collins J, Mackay H, Isenring E, Marshall S. Is telehealth effective in managing malnutrition in community-dwelling older adults? A systematic review and meta-analysis. Maturitas. 2018 May;111:31-46. doi: 10.1016/j.maturitas.2018.02.012. Epub 2018 Feb 20. PMID 29673830
- [Background] Chiu CJ, Kuo SE, Lin DC. Technology-embedded health education on nutrition for middle-aged and older adults living in the community. Glob Health Promot. 2019 Sep;26(3):80-87. doi: 10.1177/1757975917732351. Epub 2017 Nov 3. PMID 29099337
- [Background] Seifert A. The Digital Exclusion of Older Adults during the COVID-19 Pandemic. J Gerontol Soc Work. 2020 Aug-Oct;63(6-7):674-676. doi: 10.1080/01634372.2020.1764687. Epub 2020 May 13. No abstract available. PMID 32401181
- [Background] Yoon H, Jang Y, Vaughan PW, Garcia M. Older Adults' Internet Use for Health Information: Digital Divide by Race/Ethnicity and Socioeconomic Status. J Appl Gerontol. 2020 Jan;39(1):105-110. doi: 10.1177/0733464818770772. Epub 2018 Apr 16. PMID 29661052
- [Background] Choi NG, Dinitto DM. The digital divide among low-income homebound older adults: Internet use patterns, eHealth literacy, and attitudes toward computer/Internet use. J Med Internet Res. 2013 May 2;15(5):e93. doi: 10.2196/jmir.2645. PMID 23639979
- [Background] Mdege ND, Man MS, Taylor Nee Brown CA, Torgerson DJ. Systematic review of stepped wedge cluster randomized trials shows that design is particularly used to evaluate interventions during routine implementation. J Clin Epidemiol. 2011 Sep;64(9):936-48. doi: 10.1016/j.jclinepi.2010.12.003. Epub 2011 Mar 16. PMID 21411284
- [Background] Takemoto M, Manini TM, Rosenberg DE, Lazar A, Zlatar ZZ, Das SK, Kerr J. Diet and Activity Assessments and Interventions Using Technology in Older Adults. Am J Prev Med. 2018 Oct;55(4):e105-e115. doi: 10.1016/j.amepre.2018.06.005. PMID 30241621
- [Background] MacNab L, Francis SL, Lofgren I, Violette C, Shelley MC, Delmonico M, Xu F. Factors Influencing Dietary Intake Frequencies and Nutritional Risk among Community-Residing Older Adults. J Nutr Gerontol Geriatr. 2018 Jul-Dec;37(3-4):255-268. doi: 10.1080/21551197.2018.1524809. Epub 2018 Oct 30. PMID 30376443
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031
- [Background] Perracini MR, Mello M, de Oliveira Maximo R, Bilton TL, Ferriolli E, Lustosa LP, da Silva Alexandre T. Diagnostic Accuracy of the Short Physical Performance Battery for Detecting Frailty in Older People. Phys Ther. 2020 Jan 23;100(1):90-98. doi: 10.1093/ptj/pzz154. PMID 31612228
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Lee CC, Czaja SJ, Moxley JH, Sharit J, Boot WR, Charness N, Rogers WA. Attitudes Toward Computers Across Adulthood From 1994 to 2013. Gerontologist. 2019 Jan 9;59(1):22-33. doi: 10.1093/geront/gny081. PMID 29982458
- [Background] Jay GM, Willis SL. Influence of direct computer experience on older adults' attitudes toward computers. J Gerontol. 1992 Jul;47(4):P250-7. doi: 10.1093/geronj/47.4.p250. PMID 1624702
- [Background] Kasper JD, Freedman VA. Findings from the 1st round of the National Health and Aging Trends Study (NHATS): introduction to a special issue. J Gerontol B Psychol Sci Soc Sci. 2014 Nov;69 Suppl 1:S1-7. doi: 10.1093/geronb/gbu125. No abstract available. PMID 25342818
- [Background] Levine DM, Lipsitz SR, Linder JA. Trends in Seniors' Use of Digital Health Technology in the United States, 2011-2014. JAMA. 2016 Aug 2;316(5):538-40. doi: 10.1001/jama.2016.9124. No abstract available. PMID 27483069
- [Background] Cornwell EY, Waite LJ. Measuring social isolation among older adults using multiple indicators from the NSHAP study. J Gerontol B Psychol Sci Soc Sci. 2009 Nov;64 Suppl 1(Suppl 1):i38-46. doi: 10.1093/geronb/gbp037. Epub 2009 Jun 9. PMID 19508982
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Soysal P, Veronese N, Arik F, Kalan U, Smith L, Isik AT. Mini Nutritional Assessment Scale-Short Form can be useful for frailty screening in older adults. Clin Interv Aging. 2019 Apr 17;14:693-699. doi: 10.2147/CIA.S196770. eCollection 2019. PMID 31118593
- [Background] Hamirudin AH, Charlton K, Walton K. Outcomes related to nutrition screening in community living older adults: A systematic literature review. Arch Gerontol Geriatr. 2016 Jan-Feb;62:9-25. doi: 10.1016/j.archger.2015.09.007. Epub 2015 Sep 28. PMID 26444749
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- See also: Status of Poverty in San Antonio 2019 — http://www.sanantonio.gov/Portals/0/Files/HumanServices/FaithBased/2019PovertyReport.pdf
- See also: Food Insecurity Among Older Adults — http://www.aarp.org/content/dam/aarp/aarp_foundation/2015-PDFs/AF-Food-Insecurity-2015Update-Final-Report.pdf
- See also: 7 Facts about Older Adults and SNAP. National Council on Aging. — http://www.ncoa.org/article/7-facts-about-older-adults-and-snap